CLINICAL TRIAL: NCT02248298
Title: Efficacy of Ablative Fractional Laser-assisted Photodynamic Therapy With Short Incubation Time for the Treatment of Facial and Scalp Actinic Keratosis: 12-month Follow-up Results of a Randomized, Prospective, Comparative Trial
Brief Title: Efficacy of AFL-assisted PDT With Short Incubation Time in Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Song Ki-Hoon, Associate Professor, Dong-A University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DAUderma-04
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Actinic Keratosis
Keywords: Ablative fractional laser; Actinic keratosis; Efficacy; Photodynamic therapy; Short incubation time
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2h-AFL-PDT (Experimental): All 440 AK lesions of the 93 patients were randomly assigned to treatment with MAL-PDT (3h-MAL-PDT) or AFL-PDT with 2 hours (2h-AFL-PDT) and 3 hours (3h-AFL-PDT) of incubation time, using restricted randomization, with a computer-generated program.
  Interventions: Drug: 2h-AFL-PDT
- 3hr-AFL-PDT (Active Comparator): All 440 AK lesions of the 93 patients were randomly assigned to treatment with MAL-PDT (3h-MAL-PDT) or AFL-PDT with 2 hours (2h-AFL-PDT) and 3 hours (3h-AFL-PDT) of incubation time, using restricted randomization, with a computer-generated program.
  Interventions: Drug: 3h-AFL-PDT
- 3hr-MAL-PDT (Active Comparator): All 440 AK lesions of the 93 patients were randomly assigned to treatment with MAL-PDT (3h-MAL-PDT) or AFL-PDT with 2 hours (2h-AFL-PDT) and 3 hours (3h-AFL-PDT) of incubation time, using restricted randomization, with a computer-generated program.
  Interventions: Drug: 3hr-MAL-PDT

INTERVENTIONS:
Drug: 2h-AFL-PDT — AFL therapy was performed using a 2940-nm Er:YAG AFL (Joule; Sciton Inc., Palo Alto, CA, USA) at 300-550µm ablation depth, level 1 coagulation, 22% treatment density, and a single pulse. In the 3h-MAL-PDT group, the above mentioned procedures were not performed. Immediately after AFL treatment, an approximately 1-mm thick layer of MAL (Metvix, PhotoCure ASA, Oslo, Norway) was applied to the lesion and on 5 mm of surrounding normal tissue. The area was covered with an occlusive dressing (Tegaderm, 3M, St. Paul, MN, USA). After incubation for 2 hours, the dressing and cream were removed, and the area was cleansed with saline. The area was irradiated with a red light-emitting diode lamp (Aktilite CL 128; PhotoCure ASA, Oslo, Norway) with peak emission at 632 nm, placed 5 cm away from the skin surface and total light dose of 37 J/cm-2
  Arms: 2h-AFL-PDT
Drug: 3h-AFL-PDT — AFL therapy was performed using a 2940-nm Er:YAG AFL (Joule; Sciton Inc., Palo Alto, CA, USA) at 300-550µm ablation depth, level 1 coagulation, 22% treatment density, and a single pulse. In the 3h-MAL-PDT group, the above mentioned procedures were not performed. Immediately after AFL treatment, an approximately 1-mm thick layer of MAL (Metvix, PhotoCure ASA, Oslo, Norway) was applied to the lesion and on 5 mm of surrounding normal tissue. The area was covered with an occlusive dressing (Tegaderm, 3M, St. Paul, MN, USA). After incubation for 3 hours, the dressing and cream were removed, and the area was cleansed with saline. The area was irradiated with a red light-emitting diode lamp (Aktilite CL 128; PhotoCure ASA, Oslo, Norway) with peak emission at 632 nm, placed 5 cm away from the skin surface and total light dose of 37 J/cm-2
  Arms: 3hr-AFL-PDT
Drug: 3hr-MAL-PDT — an approximately 1-mm thick layer of MAL (Metvix, PhotoCure ASA, Oslo, Norway) was applied to the lesion and on 5 mm of surrounding normal tissue. The area was covered with an occlusive dressing (Tegaderm, 3M, St. Paul, MN, USA). After incubation for 3 hours, the dressing and cream were removed, and the area was cleansed with saline. The area was irradiated with a red light-emitting diode lamp (Aktilite CL 128; PhotoCure ASA, Oslo, Norway) with peak emission at 632 nm, placed 5 cm away from the skin surface and total light dose of 37 J/cm-2.
  Arms: 3hr-MAL-PDT

SUMMARY:
Photodynamic therapy (PDT) using methyl aminolevulinate (MAL) is an effective first-line treatment for actinic keratosis (AK). Erbium: yttrium-aluminium-garnet (Er:YAG) ablative fractional laser-assisted MAL-PDT (AFL-PDT) has shown significant benefit for the treatment of AK. However, knowledge on the optimal photosensitizer incubation time for AFL-PDT is limited

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) is widely used in the treatment of superficial skin cancer. It has an excellent cosmetic outcome, and it could be considered the first-line therapy for Actinic keratosis (AK). In PDT incubation time is required so that the photosensitizer can be converted to PpIX. The recommended treatment regimen of PDT requires a relatively long incubation time with ALA (4 hours) and MAL (3 hours) before illumination. Theoretically, ablative fractional laser (AFL) pre-treatment may facilitate the penetration and distribution of topically applied drugs, since the ablated laser holes extend into the dermis, thereby possibly acting as channels for drug uptake. However, knowledge on the optimal photosensitizer incubation time for AFL-PDT is limited. The objectives of this study were to compare the efficacy, recurrence rate, cosmetic outcome, and safety between AFL-PDT with 2 and 3hours of incubation vs. conventional MAL-PDT in patients with facial and scalp AK.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* the presence of 2-10 facial AK lesions

Exclusion Criteria:

* lactating or pregnant women
* patients with porphyria
* a known allergy to any of the constituents of the MAL cream and lidocaine
* patients with systemic disease
* history of malignant melanoma
* tendency for melasma development or keloid formation
* any AK treatment of the area in the previous 4 weeks
* any conditions associated with a risk of poor protocol compliance
* patients on immunosuppressive treatment

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Difference of the efficacy between 3h-AFL-PDT, 2hr-AFL-PDT and 3h-MAL-PDT | Efficacy was evaluated at 3 months and 12 months after treatment
  The response was classified as either complete response (complete disappearance of the lesion) or incomplete response (incomplete disappearance of the lesion)

SECONDARY OUTCOMES:
Difference of the cosmetic outcome between 3h-AFL-PDT, 2hr-AFL-PDT and 3h-MAL-PDT | Cosmetic outcome was assessed by each investigator for all lesions that achieved a complete response at 12 months
  It was graded as excellent (slight redness or pigmentation change), good (moderate redness or pigmentation change), fair (slight-to-moderate scarring, atrophy, or induration), or poor (extensive scarring, atrophy, or induration).

OTHER OUTCOMES:
Difference of the recurrence rates and safety between 3h-AFL-PDT, 2hr-AFL-PDT and 3h-MAL-PDT | within 12 months after each treatment
  If the case of complete response of lesions, all patients were reviewed at 12 months to check recurrence.
  Adverse events reported by the patient were noted at each follow-up visit, including severity, duration, and need for additional therapy. All events due to PDT were described as phototoxic reactions(e.g. erythema, burning sensation, swelling, bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-A University, Busan, Dong Dae Sin-dong, Seo-gu, South Korea

REFERENCES:
- [Derived] Choi SH, Kim KH, Song KH. Efficacy of ablative fractional laser-assisted photodynamic therapy with short-incubation time for the treatment of facial and scalp actinic keratosis: 12-month follow-up results of a randomized, prospective, comparative trial. J Eur Acad Dermatol Venereol. 2015 Aug;29(8):1598-605. doi: 10.1111/jdv.12953. Epub 2015 Feb 1. PMID 25640401